CLINICAL TRIAL: NCT04959643
Title: Systematic Screening for Viral Hepatitis B and C at the PASS Consultation of the Montpellier University Hospital
Acronym: dHEPass
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0439 -UF-8029
Record Dates: First submitted 2021-06-18; First posted 2021-07-13 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-10

CONDITIONS: Hepatitis C; Hepatitis B; Addiction
Keywords: Hepatitis; Viral hepatitis; Hepatitis B; Hepatitis C; Addiction; Rapid orientation tool; TROD; Continuous health care center; PASS
MeSH Terms: conditions — Hepatitis C; Hepatitis B; Behavior, Addictive; Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A high number of people are infected by viral hepatitises B and C without knowing it, especially vulnerable population such as the ones who come in consultation in continuous health care access center (Permanence d'accès aux soins, PASS). Now that these infections can be rapidly treated, it is essential to diagnose them the quickest possible. The Identification and Diagnostic Orientation Test (Test de repérage et d'orientation diagnostique, TROD) technique is a rapid tool allowing to screen for hepatitis B and C by a simple capillary sample.

The study aims to evaluate the accptability of a systematic screening using TROD for hepatitis B and C in adults in a PASS consultation in Montpellier.

We also want to estimate the prevalence of theses infections in the population, to describe the HBV and HCV care cascades, to evaluate the acceptability of vaccinal catch-up for HBV, and to describe people with hepatits.

DETAILED DESCRIPTION:
Context :

Even if the rate of under-screening for viral hepatitis B and C is getting better, the situation is still concerning. In France, it has been estimated that about 100 000 people have a positive serology for hepatitis C, and that 75,000 are unaware of it. People in vulnerable situations such as migrants or people in very precarious situations have an increased risk of having been infected by one of these two viral hepatitises.

The Précavir study established the effecacy of systematic screening for viral hepatitis during a consultation at a continuous health care access center (Permanence d'accès aux soins, PASS). Screening in the same location as the consultation is recommended, as well as the creation of a clear care pathway (Roudot-Thoraval et al. BEH 14-15 2017).

According to another study conducted in the Ile de France region, in consultations dedicated to migrants, the prevalences of hepatitis B and C were 6.8% and 1.8% respectively; whereas the vast majority of infected persons were unaware of their positivity (Revault et al. BEH 14-15; 2017). These vulnerable populations are a priority for individuals and for public health in terms of viral hepatitis screening, care and prevention.

Systematic screening for hepatitis C is justified by the now universal access to treatment and by the remarkable efficacy (>95%) of new treatments against the hepatitis C virus. These pan-genotypic treatments are prescribed for a short amount of time and have very few adverse effects. Systematic screening as well as the implementation of treatment against hepatitis C are essential in a view to obtain the elimination of hepatitis C in 2030 for the WHO and in 2025 for France. To this date, without screening and systematic initiation of treatment, the various models are unanimous that this objective cannot be achieved. We must therefore take advantage of all medical opportunities to offer this simple and cost-effective screening.

A double challenge resides for the hepatitis B: to offer treatment to people with chronic viral hepatitis B and to make a systematic catch-up vaccination, which also makes it possible to curb the risk of new transverse contaminations within communities or families.

As the recruitment will take place at the Montpellier PASS, the study population is said to be vulnerable, in great precariousness, and not necesseraly up to date with social coverage or administrative documents. Recruiting this population is essential because it is the target of our study, and will help them get in touch with the healthcare system. Moreover, access to screening first and then to care is a determining public health issue to improve the health of this population and to reach the objectives of eliminating and limiting the circulation of these viruses.

The use of the rapid identification and diagnostic orientation test (Test de repérage et d'orientation diagnostique, TROD) technique is interesting in this context because it can be deployed outside of a classic screening structure, using a simple capillary sample. This type of screening has proven its effectiveness in the diagnosis of infectious diseases in populations with difficult access, and especially in the management of HIV and hepatitis.

In addition, our acceptability study in the Montpellier PASS follows the recommendations of the health authorities as closely as possible. Indeed, the French National Authority for Health (Haute Autorité de Santé, HAS) has issued recommendations for the use of HCV and HBV screening using TROD in certain health care structures and in particular PASS (Place des tests rapides d'orientation diagnostique (TROD) dans la stratégie de dépistage de l'hépatite C, RECOMMANDATION EN SANTÉ PUBLIQUE, 27 mai 2014; Place des tests rapides d'orientation diagnostique (TROD) dans la stratégie de dépistage de l'hépatite B, RECOMMANDATION EN SANTÉ PUBLIQUE, 06 juillet 2016).

Objectives :

* The main objective is to evaluate the acceptability of the systematic hepatitis B and C screening using the TROD in adults in PASS consultations in Montpellier.
* The secondary objectives are to :

  * Determinate the seroprevalence of hepatitises B and C in our population
  * Describe the care cascade of hepatitises B and C using the test and treat model
  * Evaluate the rate of undetectable viral hepatitis C 12 weeks after the ending of the hepatitis C antiviral treatment
  * Evaluate the acceptability of the catch-up vaccination in people with a negative hepatitis B serology
  * Describe the populations with hepatitises

Methodology:

This prospective study evaluating the acceptability of a systematic screening procedure will include all adults coming to a PASS in Montpellier.

The study will offer them a rapid screening of hepatitises B and C using the TROD. This is recommended by the national authorities and actually offered at PASS in Montpellier but not in the same location, which creates a large drag to systematic screening. Participants would have the screening in situ, and the results immediately.

We will evaluate the rate of performed TROD out of the number of people to whom the TROD have been offered.

Recruiting 600 participants will allow us to estimate a screening acceptabity of 80% with a +/- 3.2% precision. This will allow us to estimate an expected VHC prevalence of 5% with a +/-2.5% precision. If 30 participants have a chronic hepatitis, we will estimate an expected rate of 80% efficacively treated patients at 3 months with an 95% confidence interval of 66% to 90%.

Regarding the analyses, we will first describe the sociodemographic caracteristics of the participants. Chronic HBV and HCV infections will be described with their 95% condidence interval. The number of people in the care cascades will be calculated. Finally, the rate of therapeutic success 12 weeks after the ending of the antiviral hepatitis C treatment will be calculated and factors associated to therapeutic success for HBV or HCV will be analysed in univariate or multivariate models if the number of treatment failures allows it.

Program :

In the inclusion visit, an explaination of benefits of hepatitis screening and the study will be offered. The non-objection to partipation will be noted. A simple questionnaire will be completed by the nurse, with information already collected for usual care.

If the TROD is positive : immediate consultation with a hepatologist or a general practitioner from the addictology service, clinical examination, somatic complication of addiction, confirmation of HBV or HCV by blood sample, eventual pre-therapeutic assessment for chronic hepatitis B and or C. Participants will be invited to come back 7 days later. A social assistant will work to open the participant's rights to an healthcare.

If the TROD are negative : offering a hepatitis B cath-up vaccination, end of participation.

For non-included patients : age, sex and reason of non participation will be collected if the patient don't object.

- First follow up visit (D7 +/-3 days) If positive viral HBV ADN : medical examination, results announcement, prescription for an antiviral treatment, counselling, evaluation of risk practices, next consultation proposed in 3 months.

If active chonic hepatitis C : medical examination, prescription for an antiviral pangenotypic treatment, counselling, evaluation of risk practices, next consultation proposed in 2 or 3 months depending of the treatment.

- Second follow up visit (HBV : W12 +/- 10 days; HCV : W8 +/- 3 days or W12 +/- 10 days) If treated B hepatitis (W12) : medical examination, evaluation of medication adherence, drug tolerance, blood sample, new prescription if needed, counselling, risk practices evalueation, participation in the will be over but the patient will have a regular medical follow up.

If treated C hepatitis (2 or 3 months) : medical examination, medical adherence evaluation, drug tolerance evaluation, risk practices evaluation, counselling, next follow-up visit given : 12 weeks after the treatment ending.

Third follow up visit Hepatitis C : 12 weeks after the treatment ending : medical examination, drug tolerance evaluation, blood sample, risk practices evaluation, counselling, healing announcement 7 days later by phone or new consultation depending of the participant's will. End of the study.

Feasability:

The PASS have a translation software use routinely to communicate with non French speaking population. A simple and clear information notice has been created to ease the comprehension.

A pratical formation to use the TROD will be given to the PASS nurse before the study.

The number of patients seen at the PASS in 2019 was 1,110 meaning 20 consultation per workday : we can guess that we will be able to include 40 patients a week and 600 patients a year.

ELIGIBILITY:
Inclusion Criteria:

* People of 18 years old and more
* Non objection to be a participant of the study

Exclusion Criteria:

* Exclusion period determined by a previous study
* Judicial protection (sauvegarde de justice, tutelle or curatelle)
* Impossibility of offering clear information to the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults in Montpellier's PASS consultation
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Rate of performed TROD | Inclusion visit
  Proportion of performed TROD out on the number of people it has been offered.

SECONDARY OUTCOMES:
Prevalence of hepatits B in the population | Inclusion visit
  Number of positive TROD for hepatitis B out on the number of people with a performed TROD
Prevalence of hepatits C in the population | Inclusion visit
  Number of positive TROD for hepatitis C out on the number of people with a performed TROD.
Care Cascade for HBV | 3 months
  Number of people with positive AgHBs, number of AgHBs+ people knowing their status, number fo AgHBs+ people treated, number of AgHBs+ people treated with an indetectable viral load or significative diminution
Care Cascade for HCV | 6 months
  Number of people with TROD VHC+, number of people knowing their VHC+ status, number of people with VHC ARN, number of treated people with VHC ARN, Numberof people with undetectable VHC ARN 12 weeks after the hepatitis antiviral treatment ending related to the number of people treated with hepatitis C antiviral treatment.
Age | Inclusion visit
  Year of birth is collected. Age is calculed as the difference between the the year of inclusion visit and the year of birth.the serological status, actual medication.
Sex | Inclusion visit
  Male, Female or undetermined.
Social care access | Inclusion visit
  Access to social care is asked : Yes/No. If yes, the participant can precise his social security and complementary health insurance statuses.
Housing status | Inclusion visit
  Permanent housing/ Temporary housing / Homelessness asked by the investigator..
Life location in the last 6 months | Inclusion visit
  France / Eastern Europe / Russia and ex-USSR / Africa (multiple answers possible).
Smoking status of people | Inclusion visit
  Non-smoker / Former smoker / Actual smoker.
Alcohol high use | Inclusion visit
  More than 10 glasses a week : Yes/no.
Usage of a care facility in Montpellier in the last year | Inclusion visit
  Yes/No.
Knowing of the serological status | Inclusion visit
  Last known serological status for hepatitis B
Knowing of the serological status | Inclusion visit
  Last known serological status for hepatitis C.
Weight of people with hepatitis | Inclusion visit
  Weight in kilograms.
Height of people with hepatitis | Inclusion visit
  Height in centimeters.
Cardiac frequency of people with hepatitis. | Inclusion visit
  In beats per minutes.
Blood pressure of people with hepatitis | Inclusion visit
  Systolic blood pressure measured in mmHg.
Blood pressure of people with hepatitis | Inclusion visit
  Diastolic blood pressure measured in mmHg.
Signs of hepatocellular insuffisance of people with hepatitis. | Inclusion visit
  Yes/No. Determined by the investigator.
Signs of portal hyperpressure of people with hepatitis. | Inclusion visit
  Yes/No. Determined by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Helene DONNADIEU RIGOLE, MH PD, Principal Investigator — Biochemistry department
Locations (1):
- CHU Montpellier, St Eloi Hospital,, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: No